CLINICAL TRIAL: NCT01414439
Title: Group Psychotherapy Among Congestive Heart Failure Patients as a Way to Reduce Psychological Distress and Increase Psycho-social Adjustment
Brief Title: Group Psychotherapy Among Congestive Heart Failure Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: MMC-chf
Record Dates: First submitted 2011-05-02; First posted 2011-08-11 (Estimated); Last update posted 2011-08-30 (Estimated); Status verified 2011-08

CONDITIONS: Congestive Heart Failure (CHF)
MeSH Terms: conditions — Heart Failure | interventions — Psychotherapy, Group

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Congestive Heart Failure Patients: 40 patients diagnosed with heart failure at levels III and IV, according to the classification of the NYHA will participate in the research. The researchers will randomly allocate the patients to the treatment group or the control group. The subjects in the treatment group will participate in Existential Group Therapy, while the subjects in the control group will not participate in the treatment until after the completion of the study. Psychological data will be collected in the form of a self-reported questionnaire completed by all participants prior to the beginning of the research and again upon completion of the final group session.
  Interventions: Behavioral: Existential Group Therapy

INTERVENTIONS:
Behavioral: Existential Group Therapy — The treatment will be given in two groups of eight to ten participants each one and will consist of one hour weekly sessions over a period of seven weeks. Dividing the subjects into small groups allows reference to all members of the group. The group facilitators will be two psychologists who work in co therapy.
  Other Names: group therapy; Supportive-Expressive Group Therapy

SUMMARY:
This study will examine the efficacy of group therapy utilizing the Existential Approach in heart failure patients when compared to a control group of patients who are waiting for the same group treatment. This comparison will be achieved by measuring changes in the variables studied namely, the levels of psychological distress and levels of psycho-social adjustment.

DETAILED DESCRIPTION:
Among all medical conditions, patients with heart failure report significantly poorer quality of life than do the other patients (1). The existing literature describes a wide range of negative emotions common among patients with heart failure; these include everything from depression, anxiety, submission and helplessness to a profound sense of "discord and brokenness." The prevalence of depression, ranging from 11% to 25% among heart disease outpatients and 35% to 70% among those who are hospitalized (2). By comparison, the overall percentage of the population suffering from depression is about 6.6%. Psychological depression appears to be an important predictor of rehospitalization among persons who have been admitted with coronary artery disease (3). In addition, depression in patients with heart failure was found to be associated with the course of the disease and its prognosis. For example, it was found that in patients with heart failure, a diagnosis of Major Depression was correlated with a higher rate of mortality (4), and depressive symptoms predicted short-term worsening of heart failure symptoms (5). The reduction in quality of life that was also found to be common in patients with heart failure is also a prognostic factor for repeated hospitalizations and death (6).

The high prevalence of distress among the population of patients with heart failure, along with the broad impact on the patient's quality of life, requires attention to detail and the implementation of interventions aimed at reducing levels of distress. Very few studies describe interventions aimed at alleviating distress in patients with heart failure. Cognitive Behavioral Therapy is reported to improve both the functional and emotional levels of these patients, resulting in the relief of their symptoms of depression. Using relaxation, Bio-Feedback devices have also achieved a reduction in depression of heart failure patients. Research testing the efficacy of psychological treatment using the interpersonal approach now is being performed; it is funded by the U.S. NIMH and is, at present, in the initial recruitment stages (National Institute of Mental Health, 2010). Studies examining the beneficial effects of group therapy are few in number and most of them utilize a Cognitive Behavioral approach. This therapeutic orientation has been found to be effective when the disease is moderate or the prognosis is favorable. However, outcomes tend to differ greatly when it comes to patients in advanced stages of the condition. These patients are also confronted with fundamental aspects of their own mortality. A large body of literature about psychological interventions for these patients exists. Many of these interventions are based on an Existential Approach aimed at facilitating responses to the unique distress of patients in an advanced stage of the disease (7).

This study examines the contribution of a group therapy program based on the Existential Approach aimed at reducing distress in patients with heart failure.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of heart failure at levels III and IV, according to the classification of the NYHA (New York Heart Association) for 3 months or more.
* Clinical diagnosis of LVEF less than 50% or were on diuretic therapy for more than three months with at least one previous hospitalization due to heart failure disease.

Exclusion Criteria:

* uncertain prognosis for 12 months due to other conditions.
* acute coronary disease in recent months.
* existence of another life-threatening illness of the patient (such as active cancer, chronic kidney failure).
* severe neurological problem (Brain syndrome / orientation problem/ difficult peripheral neuropathy).
* severe mental illness (active psychosis / suicide risk / severe dementia).
* linguistic limitations (such as misunderstanding of the Hebrew language / stuttering / untreated audio impairment).
* a significant functional problem (such as unconsciousness / connection to respiration device / confined to a wheelchair or bed / severe walking disability / needs help with complete basic daily activities).
* objective limit that endangers liability for participation in the seven meetings (such as remote residential / tourist / convict / drug addict).
* subjects whose mother tongue is not Hebrew.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients diagnosed with heart failure disorder at levels III and IV
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2011-08; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Symptoms of Emotional Distress | an expected average of 7 weeks.
  Symptoms of Emotional Distress: The BSI questionnaire (The Brief Symptom Inventory), measuring levels of depression, anxiety and somatization of the subject, will be used.

SECONDARY OUTCOMES:
Patients' Psychosocial adjustment | an expected average of 7 weeks.
  Patients' Psychosocial adjustment: The PAIS-SR questionnaire (Psychological Adjustment to Illness Scale-Self Report), will be used. This questionnaire reflects the patient's adjustment in such areas as employment and leisure activities.

CONTACTS AND LOCATIONS:
Overall Officials: Morris Mosseri, Professor, Principal Investigator — Department of Cardiology, Meir Medical Center, Israel
Locations (1):
- : Department of Cardiology, Meir Medical Center, Kfar Saba, Israel

REFERENCES:
- [Result] Juenger J, Schellberg D, Kraemer S, Haunstetter A, Zugck C, Herzog W, Haass M. Health related quality of life in patients with congestive heart failure: comparison with other chronic diseases and relation to functional variables. Heart. 2002 Mar;87(3):235-41. doi: 10.1136/heart.87.3.235. PMID 11847161
- [Result] O'Connor CM, Joynt KE. Depression: are we ignoring an important comorbidity in heart failure? J Am Coll Cardiol. 2004 May 5;43(9):1550-2. doi: 10.1016/j.jacc.2004.02.003. No abstract available. PMID 15120810
- [Result] Levine JB, Covino NA, Slack WV, Safran C, Safran DB, Boro JE, Davis RB, Buchanan GM, Gervino EV. Psychological predictors of subsequent medical care among patients hospitalized with cardiac disease. J Cardiopulm Rehabil. 1996 Mar-Apr;16(2):109-16. doi: 10.1097/00008483-199603000-00005. PMID 8681155
- [Result] Jiang W, Alexander J, Christopher E, Kuchibhatla M, Gaulden LH, Cuffe MS, Blazing MA, Davenport C, Califf RM, Krishnan RR, O'Connor CM. Relationship of depression to increased risk of mortality and rehospitalization in patients with congestive heart failure. Arch Intern Med. 2001 Aug 13-27;161(15):1849-56. doi: 10.1001/archinte.161.15.1849. PMID 11493126
- [Result] Rumsfeld JS, Havranek E, Masoudi FA, Peterson ED, Jones P, Tooley JF, Krumholz HM, Spertus JA; Cardiovascular Outcomes Research Consortium. Depressive symptoms are the strongest predictors of short-term declines in health status in patients with heart failure. J Am Coll Cardiol. 2003 Nov 19;42(10):1811-7. doi: 10.1016/j.jacc.2003.07.013. PMID 14642693
- [Result] Konstam V, Salem D, Pouleur H, Kostis J, Gorkin L, Shumaker S, Mottard I, Woods P, Konstam MA, Yusuf S. Baseline quality of life as a predictor of mortality and hospitalization in 5,025 patients with congestive heart failure. SOLVD Investigations. Studies of Left Ventricular Dysfunction Investigators. Am J Cardiol. 1996 Oct 15;78(8):890-5. doi: 10.1016/s0002-9149(96)00463-8. PMID 8888661
- [Result] Spiegel D, Classen C. Group therapy for cancer patients. A research-based handbook of psychosocial care. New York: Basic, 2000.